CLINICAL TRIAL: NCT01117909
Title: Effects of Talocrural Joint Mobilizations in the Treatment of Subacute Lateral Ankle Sprains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Dr. Terry Grindstaff, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14919
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Ankle Sprain
Keywords: ankle sprain; athletic injury; arthritis
MeSH Terms: conditions — Ankle Injuries; Athletic Injuries; Arthritis | interventions — Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Laying of hands" plus standard therapy (Sham Comparator): Subjects will lie on their back as if they were receiving the joint mobilization treatment and the therapist will place their hands in a position as if to perform the mobilization but no movement will occur. Standard therapy will consist of ankle strengthening exercises with elastic bands, balance, active ROM, and 20 minutes of ice bag application, elevation and compression
  Interventions: Other: Sham intervention
- Standard therapy with joint mobilization (Experimental): This group will receive three 60-second bouts of posterior joint mobilizations applied to the ankle joint during each treatment session, in addition to standard therapy. Standard therapy will consist of ankle strengthening exercises with elastic bands, balance, active ROM, and 20 minutes of ice bag application, elevation and compression
  Interventions: Other: Mobilization therapy in addition to standard therapy

INTERVENTIONS:
Other: Mobilization therapy in addition to standard therapy — Subject will receive three 60-second bouts of posterior joint mobilizations applied to the ankle joint during each treatment session. Standard therapy will consist of ankle strengthening exercises with elastic bands, balance, active ROM, and 20 minutes of ice bag application, elevation and compression.
  Arms: Standard therapy with joint mobilization
Other: Sham intervention — Physical therapist will lay hands as if to perform the joint mobilization but no movement will occur.
  Arms: "Laying of hands" plus standard therapy

SUMMARY:
The goal is to determine if standard therapy including joint mobilizations of the ankle performed 3 times per week for 2 weeks will increase self-reported function and decrease pain in patients with mild lateral ankle sprains.

DETAILED DESCRIPTION:
The purpose of this protocol is to assess the effects of grade IV anterior to posterior joint mobilization on self-reported function, dorsiflexion range of motion and talar glide on subjects suffering from lateral ankle sprain in the past 2-10 days and exhibit 5 degree dorsiflexion deficit in range of motion or a restriction in posterior glide of the talus.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete tear of lateral ligaments with mild laxity as measured by anterior drawer test and talar tilt
* Slight reduction in function
* Anterolateral ankle tenderness
* Dorsiflexion ROM asymmetry greater than 5° compared to uninvolved limb
* Posterior talar glide restriction greater than 5° compared to uninvolved limb; or
* Posterior talar glide less than 19°, which is one standard deviation (7°) from our previously established normative values (26°)9, 10
* Suffered from grade 1 or 2 lateral ankle sprain within the last 48hr - 8 days

Exclusion Criteria:

* A history of ankle surgery that involves intra-articular fixation,
* Syndesmotic ankle sprain (to be ruled out based on clinical examination),
* History or signs of reflex sympathetic dystrophy,
* Have received manual therapy for the ankle sprain prior to enrollment
* Grade III ankle sprain.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported function | Baseline and four weeks
  We hypothesize that the group that receives joint mobilization in addition to standard therapy will show greater improvements in Functional Ankle and Ability Measure (FAAM) and FAAM-Sport (FAAM-S) scores than those who receive standard therapy alone.
Change in self-reported pain | Baseline and 4 weeks
  We hypothesize visual analog scale (VAS) scores for pain will have a greater improvement in those who received joint mobilization in addition to standard therapy when compared to standard therapy alone.

SECONDARY OUTCOMES:
Change in ankle dorsiflexion range of motion | Baseline and 4 weeks
  We hypothesize that mobilization when applied to the talocrural joint in addition to standard therapy will result in a greater increase of ankle dorsiflexion ROM than just standard therapy alone.
Change in ligamentous laxity | Baseline and 4 weeks
  We hypothesize that ligamentous laxity in both groups will be reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Grindstaff, PhD, DPT, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States